CLINICAL TRIAL: NCT05126836
Title: Cilostazol for HFpEF (Heart Failure With a Preserved Ejection Fraction)
Brief Title: Cilostazol for HFpEF
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CV-2020-29436
Record Dates: First submitted 2021-11-01; First posted 2021-11-19 (Actual); Results first posted 2023-12-15 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-11

CONDITIONS: Heart Failure With Preserved Ejection Fraction
MeSH Terms: interventions — Cilostazol

STUDY DESIGN:
Intervention Model Description: n-of-1 design
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cilostazol (Other): First week, Cilostazol 100mg twice a day
  Second week, Placebo twice a day
  Third week, Cilostazol 100mg twice a day
  Forth week, Placebo twice a day
  Interventions: Drug: Cilostazol 100Mg Tab; Drug: Placebo
- Placebo (Other): First week, Placebo twice a day
  Second week, Cilostazol 100mg twice a day
  Third week, Placebo twice a day
  Forth week, Cilostazol 100mg twice a day
  Interventions: Drug: Cilostazol 100Mg Tab; Drug: Placebo

INTERVENTIONS:
Drug: Cilostazol 100Mg Tab — Cilostazol Twice a Day
Drug: Placebo — Placebo

SUMMARY:
Determine if cilostazol improves symptoms and NTproBNP levels (heart failure blood marker) in heart failure with preserved ejection fraction (HFpEF) - a prevalent syndrome without targeted evidence-based treatment.

This will be assessed in a prospective 1-month single blinded study with 2 cross-overs n-of-1 study design with placebo and cilostazol

DETAILED DESCRIPTION:
Heart failure (HF) is the #1 reason for hospital admissions. About half of the patients with HF have a preserved ejection fraction (HFpEF). There is no targeted evidence-based treatment for HFpEF. We recently reported that elevating the heart rate with pacemakers conveys clinical benefits e.g. reduction in heart failure symptoms, lowering filling pressures and an increase in walk distance. Cilostazol is a PDE3 inhibitor that increases the heart rate by about 5-8 beats per minute and has other potentially beneficial HFpEF effects such as peripheral vasodilation, lusitropic effects and dromotropic effects. By activating proteinkinase A, cilostazol may also phosphorylate titin, which may reduce myocardial stiffness.

n-of-1 study design using the standard dose cilostazol formulation of 100mg twice a day approved for peripheral vascular disease. The investigators and patients are blinded. The patients serve as their own controls with two crossovers (Week 1: cilostazol or placebo - Week 2: placebo or cilostazol - Week 3: cilostazol or placebo - Week 4: placebo or cilostazol).

ELIGIBILITY:
Inclusion Criteria:

* >18 yrs
* LVEF ≥ 50% (on last assessment, <2 years)
* Diagnosis of HFpEF or Shortness of breath with NYHA Class ≥ 2 and one of the following:

  1. pulmonary edema on chest imaging or documented on exam or on loop diuretics
  2. NTproBNP >400 ng/ml in the last 24 months
  3. HFpEF>50% hospitalization in the last 3 years
  4. Qualitative echo: > mild diastolic dysfunction on echo report and > mild left ventricular hypertrophy and left atrial dilation or quantitative echo: left ventricular hypertrophy [men ≥115 g/m², women ≥95 g/m² or relative wall thickness >0.42 or any LV wall thickness >1.2cm and has LA dilation (>28ml/m2)

Exclusion Criteria:

* <18yo
* resting heart rate >100/min
* patients with LVEF <50%
* advanced end-stage heart failure,
* symptomatic COPD on home O2,
* uncontrolled severe HTN (SBP >160/100 mmHg)
* patients with life expectancy <6 months,
* end-stage liver cirrhosis,
* more than moderate valve disease,
* infiltrative myocardial disease
* constrictive pericarditis or myocarditis,
* patients unable to participate in follow up,
* pregnant patients or patients without reliable contraceptive agent for the duration of study participation),
* left ventricular outflow tract obstruction,
* bleeding dyscrasias, blood dyscrasias,
* Patients on oral ketoconazole, itraconazole, fluconazole, miconazole, fluvoxamine, fluoxetine, nefazodone, sertraline, erythromycin, clarithromycin or azithromycin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-07-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- M Health Fairview, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Aiad N, du Fay de Lavallaz J, Zhang MJ, Chaikijurajai T, Ye B, Nijjar PS, Lahiri JA, Martin CM, Alexy T, Meyer M. Cilostazol in patients with heart failure and preserved ejection fraction-The CLIP-HFpEF trial. ESC Heart Fail. 2025 Apr;12(2):1437-1446. doi: 10.1002/ehf2.15162. Epub 2024 Nov 17. PMID 39552153

RESULTS

PARTICIPANT FLOW:
Groups:
- Cilostazol First (1 Week), Then Placebo (1 Week): First week, Cilostazol 100mg twice a day
  Second week, Placebo twice a day
  Third week, Cilostazol 100mg twice a day
  Forth week, Placebo twice a day
  Cilostazol 100Mg Tab: Cilostazol Twice a Day
  Placebo: Placebo
- Placebo First, Then Cilostazol: First week, Placebo twice a day
  Second week, Cilostazol 100mg twice a day
  Third week, Placebo twice a day
  Forth week, Cilostazol 100mg twice a day
  Cilostazol 100Mg Tab: Cilostazol Twice a Day
  Placebo: Placebo
Period: Overall Study
Arm/Group | Cilostazol First (1 Week), Then Placebo (1 Week) | Placebo First, Then Cilostazol
Started | 12 | 13
Completed | 11 | 12
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Cilostazol First, Then Placebo: First week, Cilostazol 100mg twice a day
  Second week, Placebo twice a day
  Third week, Cilostazol 100mg twice a day
  Forth week, Placebo twice a day
  Cilostazol 100Mg Tab: Cilostazol Twice a Day
  Placebo: Placebo
- Total: Total of all reporting groups
Arm/Group | Cilostazol First, Then Placebo | Placebo First, Then Cilostazol | Total
Number analyzed (Participants) | 11 | 12 | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 11 | 12 | 23
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 7 | 12
  Male | 6 | 5 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 10 | 10 | 20
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: KCCQ-12
Description: The Kansas City Cardiomyopathy Questionnaire contains 12 items that measure the effect of heart failure on health and quality of life. Total scores are scaled from 0 to 100 and frequently summarized in 25-point ranges, where scores represent health status as follows: 0 to 24: very poor to poor; 25 to 49: poor to fair; 50 to 74: fair to good; and 75 to 100: good to excellent
Time Frame: 4 weeks
Measure: Median (Inter-Quartile Range); unit: units on a scale
Groups:
- Cilostazol: First week, Cilostazol 100mg twice a day
  Second week, Placebo twice a day
  Third week, Cilostazol 100mg twice a day
  Forth week, Placebo twice a day
  Cilostazol 100Mg Tab: Cilostazol Twice a Day
  Placebo: Placebo
- Placebo: First week, Placebo twice a day
  Second week, Cilostazol 100mg twice a day
  Third week, Placebo twice a day
  Forth week, Cilostazol 100mg twice a day
  Cilostazol 100Mg Tab: Cilostazol Twice a Day
  Placebo: Placebo
Arm/Group | Cilostazol | Placebo
Number analyzed (Participants) | 23 | 23
units on a scale | 47 [32 to 52] | 39 [29 to 48]

2. Secondary Outcome: NTproBNP
Description: Blood marker of heart failure severity [pg/mL], average of 2 time points 1st and 3rd week
Time Frame: 1st and 3rd week
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Cilostazol | Placebo
Number analyzed (Participants) | 23 | 23
pg/mL | 375 [68 to 974] | 448 [154 to 1056]

ADVERSE EVENTS:
Time Frame: 1 month
Description: Data on non-serious adverse events was not collected
Arm/Group | Cilostazol | Placebo
All-Cause Mortality (participants affected / at risk) | 3/23 | 5/23
Serious Adverse Events (participants affected / at risk) | 3/23 | 5/23
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cilostazol (N=23) | Placebo (N=23)
Headache (General disorders) | 3 (3) | 2 (2)
Nausea (General disorders) | 3 (3) | 1 (1)
dizziness (General disorders) | 1 (1) | 0 (0)
edema (General disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-05-16): https://cdn.clinicaltrials.gov/large-docs/36/NCT05126836/Prot_SAP_000.pdf
  • Informed Consent Form (2021-05-16): https://cdn.clinicaltrials.gov/large-docs/36/NCT05126836/ICF_001.pdf